CLINICAL TRIAL: NCT07233369
Title: Myofascial Release
Brief Title: Effect of Myofascial Release on Pain, Grip Strength, Manual Dexterity, and Quality of Life in Late-Term Rehabilitation of Hand Flexor Tendon Repairs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba Çevik, physiotherapy, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/092
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hand Flexor Tendon; Facial Mobilization; Exercise
Keywords: hand flexor tendon; facial mobilization; Exercise; pain; grip strenght; hand skills; quality of life
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: Participants were divided in two groups. One group will get intervention. One group will be the control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial mobilization group (Experimental): This group will get a specific programme that combinated with conventional physiotherapy and myofascial release therapy
  Interventions: Other: Fascial mobilization therapy
- Control group (Active Comparator): This group will get conventional physiotherapy that is include range of motion exercises, electrotherapy and resistance exercise training.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Fascial mobilization therapy — Patients in this group will receive training in myofascial release exercises in addition to the exercises in the control group. Similar to the control group, patients in this group will be asked to continue home exercises five times a week for eight weeks after their two-week treatment.The patients in the study group will receive the same treatment, twice a week for 12 weeks, with each session lasting 45 minutes.
  Arms: Fascial mobilization group
Other: conventional physiotherapy — Conservative treatment methods such as TENS, Hotpack and normal joint range of motion exercises and tendon gliding exercises and streching exercise will be applied twice a week for 12 weeks, with each session lasting 45 minutes.
  Arms: Control group

SUMMARY:
The aim of this study was to investigate the effectiveness of myofascial release exercises performed in the late period compared to classical physiotherapy training in individuals with hand flexor tendon repair.

DETAILED DESCRIPTION:
The hand is the organ we use most in our daily activities, sports activities, expressing ourselves, and performing our jobs. Flexor tendon injuries are among the most common injuries to the hand. The incidence of flexor tendon injuries is estimated at 7-14 per 100,000 people. The flexor tendon can be injured by a blunt or sharp instrument, crushed, or torn by avulsion. It is difficult for tendons to heal without surgery after an injury. Because tendons are composed of living cells and connective tissue, healing begins with cells from both inside and outside the tendon when the tendon ends are brought together. However, scar tissue that forms after surgery adheres the repaired tendons to the surrounding area, limiting movement. Therefore, rehabilitation protocols implemented to ensure proper gliding again and postoperative splinting are essential for tendon healing in tendon injuries are crucial. Tendon Rehabilitation Extension block splints should place the wrist in 30 degrees of flexion to reduce tension in flexor tendon repairs and minimize the risk of postoperative tendon rupture, with the metacarpophalangeal joints at 45-70 degrees of flexion and the interphalangeal joints held in near full extension or slight flexion (15 degrees). Sutures are removed two weeks postoperatively. Thanks to advances in biomechanics and clinical research, there is a general understanding that early therapy-guided tendon release is more beneficial than strict immobilization in efforts to achieve maximum functional recovery. Mobilization promotes intrinsic tendon healing, increases tensile strength, and improves tendon glide while reducing adhesion formation. All of this translates to optimized joint motion, fewer flexion contractures, and overall improved functional outcomes. Tendon repair rehabilitation programs are ideally structured to improve overall hand function while facilitating diverse soft tissue injuries. Flexor tendon rehabilitation protocols are broadly divided into three groups: immobilization, early passive mobilization, and early active mobilization. The selection of a rehabilitation protocol should be determined by considering factors such as the patient's age, ability to comply with treatment, and suture strength.

Current techniques in flexor tendon repair have led to advancements in rehabilitation practice, encouraging a shift from passive methods to early, controlled, and more active approaches. Optimal flexor tendon surgery and treatment outcomes depend on a patient-centered protocol rather than a strictly structured protocol.

Individuals aged 18-65 who have suffered a flexor tendon injury and have undergone related surgery, and who have no neurological symptoms in the repaired extremity will be included in the study.

Individuals who have previously undergone hand surgery for any reason other than this injury, who have a comorbid mental, physical, or neurological chronic illness, who have cognitive problems that impede communication, or who have any other problems that impede cooperation will not be included in the study. When we divided the included individuals into two groups, the control group will receive only conventional physiotherapy, while the study group will additionally receive myofascial release exercises. Pre- and post-treatment evaluations will be conducted. The aim of our randomized controlled trial was to investigate the effects of myofascial release on pain, dexterity, function, and quality of life in the late-stage rehabilitation of hand flexor tendon repairs.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 65,
* Having a hand flexor tendon injury and subsequent surgery,
* Not having a symptom of deterioration in the extremity being cared for,
* Having adequate communication skills,
* Voluntarily participating in the study.

Exclusion Criteria:

* Having had previous hand surgery for any reason other than this injury,
* Having a comorbid mental, physical, or neurological chronic illness,
* Having cognitive problems that prevent communication,
* Having any problem that prevents cooperation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The pain | through of the study, average 8 weeks
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Grip strength | through of the study, average 8 weeks
  A hand dynamometer will be used to measure patients' grip strength. Grip strength is measured with the Jamar hand dynamometer, recommended by the American Association of Hand Therapists (AETD) and whose validity and reliability have been confirmed in numerous studies. This device is considered the gold standard for measuring hand grip strength. Measurements will be taken before and after treatment, and three times, 10 seconds apart. Each measurement will be taken at the same difficulty level. Generally, the average of the three measurements will be taken.
Hand skills | through of the study, average 8 weeks
  The Nine-Hole Peg test, used to assess manual dexterity, involves patients quickly removing nine wooden pegs from a storage box, placing them in random holes, then collecting them from the holes and returning them to the storage compartment. The time is measured in seconds using a stopwatch, and anything over 20 seconds is considered a "loss of skill."
Short form SF-36 Quality of life | through of the study, average 8 weeks
  Individuals' quality of life will be assessed using short form 36 (SF-36). SF-36 is a 36-question scale consisting of physical function, physical role, emotional role, pain, vitality, general health, and mental health subscales.

SECONDARY OUTCOMES:
Upper extremity functionality | through of the study, average 8 weeks
  The Questionnaire for Arm, Shoulder, and Hand Disabilities (Q-DASH) will be used to assess individuals' upper extremity functions. This questionnaire is a self-administered measurement tool with validated validity and reliability in Turkish. The validity and reliability of the Turkish version of the DASH questionnaire (DASH-T) was conducted in Turkey by Düger et al. in 2006. The questionnaire, consisting of 30 questions, assesses the individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with a higher score indicating better outcomes.
Range of Motion | through of the study, average 8 weeks
  A Universal Goniometer will be used to assess normal range of motion. Measurements will be made regarding shoulder flexion, extension, abduction, adduction, internal and external rotation ranges of motion in three planes of the upper extremity shoulder joint, and the results will be recorded in degrees.
Kinesiophobia | through of the study, average 8 weeks
  This is the measure we will use to assess patients' fear of movement in our study. This scale, frequently used in the literature, is based on fear avoidance, fear of work-related activities, and fear of movement or re-injury.
Daily living activities | through of the study, average 8 weeks
  It is a 15-question questionnaire that measures the severity of wrist pain and the level of disability in daily life activities.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Çevik, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sheereen FJ, Sarkar B, Sahay P, Shaphe MA, Alghadir AH, Iqbal A, Ali T, Ahmad F. Comparison of Two Manual Therapy Programs, including Tendon Gliding Exercises as a Common Adjunct, While Managing the Participants with Chronic Carpal Tunnel Syndrome. Pain Res Manag. 2022 Jun 8;2022:1975803. doi: 10.1155/2022/1975803. eCollection 2022. PMID 35719196
- [Result] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Result] Ennaciri B, Mahfoud M, El Bardouni A, Berrada MS. Exceptional laceration of flexor digitorum tendons proximal to a severe palmar hand wound: a case report with literature review. Pan Afr Med J. 2015 Nov 20;22:266. doi: 10.11604/pamj.2015.22.266.7495. eCollection 2015. PMID 26958129
- [Result] Mattar TG, Junior RM, Cho AB, Paula EJ, Rezende MR. COMPARATIVE STUDY BETWEEN TRADITIONAL TENOLYSES AND WITH INTRAOPERATIVE AWAKENING PERFORMED ON THE FLEXOR OSTEOFIBROUS TUNNEL REGION OF THE HANDS (ZONE 2). Rev Bras Ortop. 2015 Dec 8;44(4):324-9. doi: 10.1016/S2255-4971(15)30161-0. eCollection 2009 Jan. PMID 27022514
- [Result] Quadlbauer S, Pezzei Ch, Jurkowitsch J, Reb P, Beer T, Leixnering M. Early Passive Movement in flexor tendon injuries of the hand. Arch Orthop Trauma Surg. 2016 Feb;136(2):285-93. doi: 10.1007/s00402-015-2362-z. Epub 2015 Dec 11. PMID 26659831
- [Result] Watanabe K, Ota H, Sasaki H. Eight-strand Cross-locked Cruciate Flexor Tendon Repair Using Double-stranded Suture: A Description of the Surgical Technique. Plast Reconstr Surg Glob Open. 2016 Nov 7;4(11):e1048. doi: 10.1097/GOX.0000000000001048. eCollection 2016 Nov. PMID 27975005
- [Result] Stevens KA, Caruso JC, Fallahi AKM, Patino JM. Flexor Tendon Lacerations. 2023 Jun 20. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493223/ PMID 29630275
- [Result] Ranjan V, Mehta M, Mehta M, Mishra P, Joshi T, Kumar T. The Outcomes of Flexor Tendon Injury Repair of the Hand: A Clinico-Epidemiological Study. Cureus. 2023 Jan 18;15(1):e33912. doi: 10.7759/cureus.33912. eCollection 2023 Jan. PMID 36819329
- [Result] Moradi A, Menendez ME, Kachooei AR, Isakov A, Ring D. Update of the Quick DASH Questionnaire to Account for Modern Technology. Hand (N Y). 2016 Dec;11(4):403-409. doi: 10.1177/1558944715628006. Epub 2016 Feb 2. PMID 28149205